CLINICAL TRIAL: NCT00573495
Title: A Study of hTERT/Survivin Multi-peptide Vaccine With Daclizumab and Prevnar for Patients With Metastatic Breast Cancer
Brief Title: Multipeptide Vaccine for Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 08107
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Breast Neoplasm; Breast Cancer; Cancer of the Breast; Carcinoma, Ductal
Keywords: Advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal | interventions — Telomerase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hTERT/Survivin Multi-Peptide Vaccine (Experimental)
  Interventions: Biological: hTERT/Survivin Multi-Peptide Vaccine

INTERVENTIONS:
Biological: hTERT/Survivin Multi-Peptide Vaccine — 100 mcg subcutaneous every 2 weeks four times, then monthly up to 28 vaccinations
  Other Names: hTERT; Telomerase

SUMMARY:
This is a study on how to activate the immune system with a vaccine. The vaccine is made up of two proteins found in breast cancer: telomerase and survivin. The vaccine is given in combination with other drugs that may also have an effect on the immune system and attack the cancer.

The goals of the study are:

1. to test the safety of the combination of agents
2. to find out what effects the treatment has on advanced breast cancer

DETAILED DESCRIPTION:
Patients with advanced breast cancer may often fail standard of care treatments for metastatic disease. This research is studying a combinations of agents that impact the immune system.

About >85% of all human cancers, including breast cancer, express telomerase (hTERT) activity. Targeting hTERT immunologically may also minimize immune escape due to antigen loss because mutation or deletion of hTERT may be incompatible with sustained tumor growth. hTERT Multi-Peptide Vaccine is made up of 1540 hTERT peptide and cryptic peptides selected for "low-affinity" binding to HLA-A2 in order to increase the likelihood that the host immune system would ignore them, and then they have been modified by changing the first amino acid of the peptides to tyrosine in order to increase HLA - A2 affinity. The two "heteroclitic" peptides are R572Y (YLFFYRKSV) and D988Y (YLQVNSLQTV), which bind HLA-A2 with high avidity and elicit specific CTL (cytotoxic T lymphocyte) responses using healthy donor mononuclear cells in vitro. In addition, in mouse models, these peptide vaccines elicit lytic CTL responses which are protective against tumor challenges using a TERT-expressing murine tumor.

Subjects will also be immunized with a peptide vaccine derived from survivin, an important anti-apoptotic protein which is overexpressed in a broad range of malignancies including breast cancer. Survivin may be an ideal and "universal" tumor antigen since it is overexpressed in a wide variety of cancers yet terminally differentiated adult cells do not express the protein.

CMV derived CTL epitopes will be used as positive control peptides.

Daclizumab is a humanized anti-human CD25 monoclonal antibody that binds specifically to CD25 expressing cells, including Treg cells, and inhibits its proliferation.

Prevnar is designed to augment T-helper cell immunity.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV breast cancer that has failed at least one conventional therapy for metastatic disease
* HLA-A2 positive
* Measurable or evaluable disease
* ECOG performance status 0-1
* Negative contrast CT or MRI scan of the brain within 30 days of treatment
* Negative pregnancy test within 14 days of treatment for women of childbearing potential

Exclusion Criteria:

* History of brain metastases within the last 4 years
* The use of chemotherapy, radiation therapy, immunosuppressive drugs, systemic glucocorticoids, growth factors, or experimental therapy, and anti-coagulants within 14 days prior to treatment
* Initiation of hormonal agent in the 30 days before treatment
* Initiation of Herceptin in the 30 days prior to treatment.
* History of bone marrow or stem cell transplantation
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-11; Primary Completion 2011-07 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety | Up to 30 days after the last vaccination

SECONDARY OUTCOMES:
Immunologic response | After 4th vaccination, then after every 3-4 vaccinations, and then every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fox, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Medical Center, Philadelphia, Pennsylvania, United States